CLINICAL TRIAL: NCT07385417
Title: Electroporation Treatment for Early AF Management in Heart Failure With Preserved Ejection Fraction (HFpEF) Pilot Study
Acronym: E-TEAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardioangiologisches Centrum Bethanien (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20221013 E-Team V.2
Record Dates: First submitted 2023-11-30; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Electroporation Treatment for Early AF Management in Heart Failure with preserved Ejection Fraction (HFpEF) Pilot Study
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AF Ablation with electroporation (Active Comparator): Patient in this arm will receive AF-Ablation
  Interventions: Procedure: AF Ablation
- best medical AF treatment including rhythm and rate control (n=100) (No Intervention): In this group patients reeive anti arrhythmia medication or ECV

INTERVENTIONS:
Procedure: AF Ablation — Atrial fibrillation ablation
  Other Names: Medication or ECV
  Arms: AF Ablation with electroporation

SUMMARY:
The proposed pilot study is a prospective, randomized, single-center feasibility study, enrolling 200 patients with symptomatic paroxysmal AF. Per protocol, 100 patients will undergo a FARAPULSE electroporation PVI and 100 patients will receive standard AF medical treatment.

Prior enrollment, all patients will be informed on the risk and benefits of the PVI procedure as well as the medical treatment. In addition, particular information on the rationale of the study, including a detailed risk/benefit analysis, will be provided to all patients.

ELIGIBILITY:
Inclusion Criteria:

1. Seeking emergency (E) treatment including emergency room (ER) presentation
2. Paroxysmal AF diagnosed according to current ESC guidelines
3. Diagnosis of HFpEF according to ESC guidelines 2021 (clinical symptoms, EF>50%, objective evidence of functional abnormality: LV diastolic dysfunction, NT-proBNP (non acute setting): sinus rhythm: 125pg/ml or AF: 365pg/ml, vs. acute HF: >450 pg/ml if aged <55 years, >900 pg/ml if aged between 55 and 75 years and >1800 pg/ml if >75ys.
4. Age between 18 and 80 years
5. Left atrial size, LA < 55mm
6. Left ventricular ejection fraction, EF >50%
7. Patients able to provide informed consent and willing to comply with all pre-, post- and follow up requirements as per study protocol -

Exclusion Criteria:

1. Currently participating in an interventional (drug, device, biologic, etc.) clinical trial
2. Any disease that limits life expectancy to less than one year
3. Contraindications for PVI
4. Contraindication for AAD therapy
5. Active systemic infection
6. Thrombocytosis, thrombocytopenia
7. Known pre-existing hemi-diaphragmatic paralysis
8. Any untreated or uncontrolled hyperthyroidism or hypothyroidism
9. Reduced immune function or otherwise at high risk for infection per physician discretion
10. Active malignancy or history of chemotherapy or radiation treatment
11. Prior left atrial ablation or surgical procedure (including left atrial appendage closures)
12. Any cardiac surgery, myocardial infarction, PCI/PTCA or coronary artery stenting which occurred within the 3 months before the eligibility assessment
13. Instable angina pectoris
14. Primary pulmonary hypertension
15. Any condition contraindicating chronic anticoagulation
16. Any cerebral ischemic event (strokes or TIAs) which occurred within the 3 months before the consent date
17. Presence of any cardiac prosthetic valves
18. Left atrial diameter > 55 mm (anteroposterior) by TTE
19. Presence of any pulmonary vein stents
20. Presence of any pre-existing pulmonary vein stenosis (identified by CT or MRI and defined as at least 70% reduction of the PV diameter)
21. Endocarditis, pericarditis or pericardial effusion
22. Pregnant or breastfeeding women or women of childbearing potential not on adequate birth control.
23. Substance abuse
24. Unwilling to follow the study protocol and to attend follow-up visits

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2026-04-12 (Estimated); Study Completion 2026-04-12 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | within the study duration of 1 Year
  composite of cardiovascular hospitalization, death, systemic embolism, stroke and emergency (E) treatment for cardiovascular reason.

SECONDARY OUTCOMES:
Secondary Endpoint | Within one year study
  major bleeding requiring intervention, phrenic nerve palsy, pericardial tamponade, thromboembolic events, atrio-esophageal fistula, death

CONTACTS AND LOCATIONS:
Overall Officials: Julian Chun, Professor, Principal Investigator — MVZ CCB
Locations (1):
- Cardioangiologisches Centrum Bethanien, Frankfurt am Main, Germany

DOCUMENTS (2):
  • Study Protocol: Version 2.1 (2025-10-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT07385417/Prot_000.pdf
  • Study Protocol: E-Team Study Protocol V2.1 (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT07385417/Prot_001.pdf